CLINICAL TRIAL: NCT01503710
Title: Early Diagnosis of Postoperative Acute Renal Failure - Using Biomarker to Predict the Outcome of Cardiac Surgery Associated Acute Kidney Injury
Brief Title: Early Diagnosis of Postoperative Acute Renal Failure-using Biomarker to Predict Outcome of Cardiac Surgery Associated Acute Kidney Injury
Acronym: NSARF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201105047RC
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-07

CONDITIONS: Acute Renal Failure; Acute Kidney Injury
Keywords: Proteinuria predict outcome; BNP and NGAL predict outcome; Pre-operative GFR and proteinuria
MeSH Terms: conditions — Acute Kidney Injury; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples are drawn before the first dialysis session after postcardiac sugary associated severe AKI ( initializing RRT). Blood is drawn into Vacutainer tubes containing EDTA, and immediately placed on ice and centrifuged within 1 h. All the samples are stored at -70°C until analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine soluble HJV could be an early diagnosis urinary biomarker of ischemia/reperfusion injury in post CPB-patients.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common syndrome on Intensive Care Unit, and renal dysfunction would result in a further morbidity and mortality. Critical ills complicated with acute kidney injury are usually accompanied with multi-organ failure. Therefore, National Taiwan University Hospital Study group of Acute Renal Failure (NSARF) realizes that the characteristics of AKI is resulted from the perfusion less of body fluid and attempt to develop therapies to prevent or attenuate AKI, which have had limited success. We attempt to use the novel biomarker soluble hemojuvelin (sHJV) to evaluate the iron homeostasis on acute kidney injury and develop new strategies and therapies such as protease inhibitors on kidney function, as safety markers to monitor toxicity and as measures of treatment effect. Besides, we will focus on validation the sensitivity and specificity of sHJV on the clinical specimen of post-operative patients from NSARF data-bank. Merge the renal function and other types of biomarkers as panel to predict the post-operative outcome. Based on the different expression of these markers, using a panel of serum and urine markers may potentially help us to distinguish between various types of insults, establish the duration and severity of injury, predict the clinical outcome and help to monitor response to treatment in AKI.

ELIGIBILITY:
Inclusion Criteria:

* AKI is defined as a serum creatinine level greater that 50% more than baseline during the first 3 postoperative days (PODs), and non-AKI, as a less than 10% increase.

Exclusion Criteria:

* Patients with chronic kidney disease (baseline estimated glomerular filtration rate < 60 mL/min/1.73 m2 as calculated by using the 4-variable Modification of Diet in Renal Disease Study equation, or protein-creatinine ratio > 100 mg/mmol) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients (cases) that developed AKI during the follow-up period of 72 h. AKI was defined as a 50% or greater increase in SCr from baseline according to the RIFLE-R criteria. For each of these cases, we then selected 20 controls from patients who also underwent open heart surgery but did not develop AKI. We matched the cases and controls as closely as possible for age, sex, baseline estimated GFR, comorbidities, medications, type of surgery and perioperative complications.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: V C Wu, M.D., Ph.D., Principal Investigator — Section of Nephrology, Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Wen-Je Ko, Taipei, Taiwan, Taiwan